CLINICAL TRIAL: NCT03176329
Title: Closed-loop Versus Conventional Ventilation Mode During Mobilization Period in Critical Care Patients : a Prospective Randomized Crossover Study
Brief Title: Closed-loop Versus Conventional Ventilation Mode During Mobilization Period in Critical Care Patients
Acronym: I-Nursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital of Melun (Other)
Responsible Party: Principal Investigator, Chelly Jonathan, MD, Hopital of Melun
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MelunH-02
Record Dates: First submitted 2017-05-28; First posted 2017-06-05 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Critical Ill Patients; Ventilated Patients
Keywords: Full closed-loop ventilation control; Critical care

STUDY DESIGN:
Intervention Model Description: Prospective randomized crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INTELLIVENT-ASV / Conventional mode (Other): Full closed-loop ventilation control (INTELLIVENT-ASV) is set 30 minutes before Nursing 1 after randomization. Ventilator is switch to conventional ventilation 30 minutes before Nursing 2
  Interventions: Other: Nursing 1 : INTELLIVENT-ASV; Other: Nursing 2 : Conventional mode
- Conventional mode / INTELLIVENT-ASV (Other): Conventional ventilation control is set 30 minutes before Nursing 1 after randomization. Ventilator is switch to full closed-loop ventilation (INTELLIVENT-ASV) 30 minutes before Nursing 2.
  Interventions: Other: Nursing 2 : INTELLIVENT-ASV; Other: Nursing 1 : Conventional mode

INTERVENTIONS:
Other: Nursing 1 : INTELLIVENT-ASV
  Arms: INTELLIVENT-ASV / Conventional mode
Other: Nursing 2 : INTELLIVENT-ASV
  Arms: Conventional mode / INTELLIVENT-ASV
Other: Nursing 1 : Conventional mode
  Arms: Conventional mode / INTELLIVENT-ASV
Other: Nursing 2 : Conventional mode
  Arms: INTELLIVENT-ASV / Conventional mode

SUMMARY:
Nursing is essential in critically ill patients care but with high risk of hypoxia, especially during mobilization. Full closed-loop control ventilation is well established for her safety in unselected ventilated critical care patients with different lung conditions compared to conventional ventilation.

The aim of this study is to assess the ability of a full closed-loop control ventilation (Intellivent-ASV, TM) to reduce hypoxia during mobilization period in unselected ventilated patients.

DETAILED DESCRIPTION:
Prospective randomized cross over study including all consecutive ventilated patient with predicted duration of ventilation > 48 hours, inspired oxygen fraction < 60% and without neuromuscular blocking agent.

Patient were randomized to be ventilated with full closed-loop control or conventional ventilation 30 minutes before the first nursing period after inclusion. The ventilator was switched in the other mode (conventional or full closed-loop respectively), 30 minutes before the following nursing period. Between this two consecutive nursing periods, ventilation mode is choosed by the attending physician.

The primary outcome was the oxygenation measured by pulse oxymetry during the nursing periods.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation for expected time >48h

Exclusion Criteria:

* Pregnancy
* Neuromuscular blocking agent (discontinuous or continuous) infusion
* Inspired oxygen fraction (FiO2) setting > or = 60%
* Mobilization contraindication (hemodynamic instability, unstable vertebral trauma, etc.)
* Neurological breathing (patients with brain injury)
* Pulse oxymetry monitoring unavailable
* Expected ventilation weaning <24h after randomization.
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Time spent with SpO2 values > 90 and < 95% | 1 day
  Pulse oxymetry monitoring

SECONDARY OUTCOMES:
Time spent with SpO2 values < or = 90% | 1 day
  Pulse oxymetry monitoring
Time spent with SpO2 values > or = 95% | 1 day
  Pulse oxymetry monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Chelly, MD, Principal Investigator — Mixed, ICU, Centre Hospitalier de Melun
Locations (1):
- Centre Hospitalier de Melun, Melun, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bialais E, Wittebole X, Vignaux L, Roeseler J, Wysocki M, Meyer J, Reychler G, Novotni D, Sottiaux T, Laterre PF, Hantson P. Closed-loop ventilation mode (IntelliVent(R)-ASV) in intensive care unit: a randomized trial. Minerva Anestesiol. 2016 Jun;82(6):657-68. Epub 2016 Mar 8. PMID 26957117
- [Background] Arnal JM, Garnero A, Novonti D, Demory D, Ducros L, Berric A, Donati S, Corno G, Jaber S, Durand-Gasselin J. Feasibility study on full closed-loop control ventilation (IntelliVent-ASV) in ICU patients with acute respiratory failure: a prospective observational comparative study. Crit Care. 2013 Sep 11;17(5):R196. doi: 10.1186/cc12890. PMID 24025234
- [Background] Clavieras N, Wysocki M, Coisel Y, Galia F, Conseil M, Chanques G, Jung B, Arnal JM, Matecki S, Molinari N, Jaber S. Prospective randomized crossover study of a new closed-loop control system versus pressure support during weaning from mechanical ventilation. Anesthesiology. 2013 Sep;119(3):631-41. doi: 10.1097/ALN.0b013e3182952608. PMID 23619172
- [Background] Arnal JM, Wysocki M, Novotni D, Demory D, Lopez R, Donati S, Granier I, Corno G, Durand-Gasselin J. Safety and efficacy of a fully closed-loop control ventilation (IntelliVent-ASV(R)) in sedated ICU patients with acute respiratory failure: a prospective randomized crossover study. Intensive Care Med. 2012 May;38(5):781-7. doi: 10.1007/s00134-012-2548-6. Epub 2012 Mar 30. PMID 22460854
- [Derived] Chelly J, Mazerand S, Jochmans S, Weyer CM, Pourcine F, Ellrodt O, Thieulot-Rolin N, Serbource-Goguel J, Sy O, Vong LVP, Monchi M. Automated vs. conventional ventilation in the ICU: a randomized controlled crossover trial comparing blood oxygen saturation during daily nursing procedures (I-NURSING). Crit Care. 2020 Jul 22;24(1):453. doi: 10.1186/s13054-020-03155-3. PMID 32698860